CLINICAL TRIAL: NCT04904432
Title: Involvement of Perilipin-1 Variants in Precocious Acute Coronary Syndrome
Brief Title: PLIN1 Variants in Precocious ACS (SCAPLIN)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-06
Record Dates: First submitted 2021-04-15; First posted 2021-05-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- young ACS patients (Other)
  Interventions: Genetic: PLIN1 gene sequencing

INTERVENTIONS:
Genetic: PLIN1 gene sequencing — One supplementary blood sample will be taken (compare to classical ACS treatment and follow up) to realize genetic analyse of PLIN1 gene, looking for mutations

SUMMARY:
This study aims to identify a genetic predisposition factor of precocious acute coronary syndrome occurrence (ACS). ACS is a major public health problem and the first cause of mortality in the world. It can be due to several risk factor such as heredity. the investigators make the hypothesis that occurrence of early ACS (defined as <50yo for men and <55yo for women) could be the initiatory event of a mild form of genetic lipodystrophy . Our previous study shown an occurrence risk of ACS about 8.3 in patients carrying a mutation in the PLIN1 gene versus patients without a mutation. The PLIN1 gene encode for perilipin 1 protein localized on the lipid droplet surface. This protein phosphorylation activates the triglycerides lipolysis. Our goals in this study are multiple: to validate the high frequency of mutations in this gene in patients with early ACS, to determine differences in triglycerides metabolism and also relapse rate between carrier and non-carrier patients of mutation in PLIN1. Our first aim will be to carry out the inclusion of 200 patients with precocious ACS. This will allow us to obtain around 15 patients carrying a mutation in the PLIN1 gene based on our previous study. the investigators will reprogramme patients' cells (carrying or not a PLIN1 mutation) in human Induce Pluripotent Stem cells (hIPSc). These hIPSc will be differentiated in cell types of interest as adipocytes or macrophages. the investigators will then study triglycerides metabolism (lipid droplet formation, localization and phosphorylation of perlipin 1) in these cells and atheroma plaque formation. Finally, the investigators will study clinical data such as relapse rate and searching for correlation with PLIN1 mutation.

ELIGIBILITY:
Inclusion Criteria:

* Age of the patient when ACS occurs (between 18 and 50yo for men, between 18 and 55yo for women)
* Written informed consent

Exclusion Criteria:

* Men <18yo or >50yo
* Women <18yo or >55yo
* ACS causes (toxic, coronary dissection)
* Congenital cardiac malformations
* Familial hypercholesterolaemia
* Pregnancy, breast-feeding women or vulnerable profile.
* Patient refusal to participate or previously included in a clinical research trial.

Ages: 10 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
PLIN1 mutation | 1 month
  sequencing PLIN1 gene to look for mutation
Lipid droplets | 3 years
  Analyze size of lipid droplets in differentiated hIPS cells

SECONDARY OUTCOMES:
relapse rate | 1 year
  Ischaemic relapse rate during the year of classical following-up

CONTACTS AND LOCATIONS:
Overall Officials: Emilie GARRIDO-PRADALIE, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France